CLINICAL TRIAL: NCT05056883
Title: A Phase III Confirmatory Study of K-237-Multi-regional, Multi-center, Placebo Controlled, Randomized, Double Blind, Parallel Group Controlled Trial in Patients With Mild COVID-19
Brief Title: A Phase III Confirmatory Study of K-237
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-237-01
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): K-237 0.3-0.4mg/kg (once daily)
  Interventions: Drug: K-237 0.3-0.4mg/kg (once daily)
- Control A (Placebo Comparator): Placebo (once daily)
  Interventions: Drug: Placebo 0.3-0.4mg/kg (once daily)

INTERVENTIONS:
Drug: K-237 0.3-0.4mg/kg (once daily) — Ivermectin 3mg tablet
  Other Names: Ivermectin 0.3-0.4mg/kg (once daily)
  Arms: Treatment A
Drug: Placebo 0.3-0.4mg/kg (once daily) — Placebo 3mg tablet
  Arms: Control A

SUMMARY:
The efficacy and safety of K-237 0.3-0.4 mg/kg orally administered once daily for 3 days will be evaluated in patients with mild COVID-19 using a randomized, double-blind, parallel-group comparative method with placebo as a control. Efficacy will be assessed using a stratified log-rank test to determine the superiority of the drug over placebo in terms of time to improvement in clinical symptoms from the start of study drug administration to 168 hours.

ELIGIBILITY:
Inclusion Criteria:

Persons who meet all of the following criteria will be eligible for this clinical trial.

1. Males and females who are 12 years of age or older at the time of obtaining consent
2. Those who are confirmed positive for SARS-CoV-2 by antigen test or RT-PCR test using specimens (nasopharynx, nasal cavity, oropharynx, or saliva) collected within 120 hours prior to obtaining consent.
3. Patients who have fevers (37.5 degrees Celsius or higher) and/or at least one of the following symptoms of Score 2 or higher at a screening test: Myalgia, sore throat, diarrhea, nausea, vomiting, cough, and shortness of breath.
4. Patients with a room air oxygen saturation (SpO2) of 96% or higher at the time of the screening test.

Exclusion Criteria:

* Subjects who meet any one of the following criteria will be excluded from this study.

  1. Patients who have had symptoms caused by COVID-19 for more than 6 days on the day of initiation of study drug administration (Day 1) with the day of onset of symptoms as Day 0.
  2. Patients who need to receive concomitant therapy or administration of prohibited drugs during the study period
  3. Patients who have taken or received drugs that have or may have antiviral activity against SARS-CoV-2 within 2 weeks prior to the start of study drug administration.
  4. Patients currently using antiviral drugs
  5. Patients with suspected complications of infectious diseases other than COVID-19
  6. Subjects with a history of COVID-19 within 1 month prior to obtaining consent
  7. Persons whose weight at the time of the screening test falls into the following categories (The first decimal place of the weight shall be rounded off.) 1) Those who are 18 years of age or older at the time of consent and weigh less than 25 kg or more than 127 kg 2) Those who are between 12 and 18 years of age and weigh less than 40 kg or 127 kg or more at the time of obtaining consent.
  8. Patients undergoing dialysis treatment
  9. Patients wno have severe liver dysfunction (hepatic dysfunction, hepatic fibrosis, etc.)
  10. Patients with poorly controlled hypertension (systolic blood pressure (SBP) of 180 mmHg or higher or diastolic blood pressure (DBP) of 110 mmHg or higher)
  11. Patients with complications of diabetic retinopathy, diabetic nephropathy, or diabetic neuropathy
  12. Patients with heart failure of NYHA Class III or higher
  13. Patients with malignant tumors or those judged to have a high possibility of recurrence
  14. Patients requiring oxygen therapy
  15. A person who has a complication of methemoglobinemia or any other disease that may cause measurement error of the pulse oximeter
  16. Patients with a history of serious drug allergy (anaphylactic shock, etc.)
  17. Pregnant women, lactating women, or women who plan to become pregnant or lactate during the study period
  18. Subjects who have had more than 400 mL of whole blood drawn within 16 weeks or more than 200 mL within 4 weeks prior to obtaining consent, or component blood (plasma and platelet components) drawn within 2 weeks
  19. Patients who have been administered IVM.
  20. Those who have participated in other clinical trials and received medication at the time of obtaining consent, or those who have received an investigational drug other than placebo for less than 16 weeks
  21. Others who are judged by the investigator or others to be inappropriate to participate in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Time from the start of study drug administration to 168 hours until the clinical symptoms reach an improving trend | Day1～11 after administration

SECONDARY OUTCOMES:
In addition to the primary endpoint, time to trend toward improvement in clinical symptoms, including headache, abdominal pain, nasal | Day1～11 after administration
Time to reach a temperature of less than 37.5 ˚C without the use of antipyretics (acetaminophen) | Day1～11 after administration

CONTACTS AND LOCATIONS:
Locations (55):
- Japan (52):
  - Hosokawa Surgical Clinic, Aichi
  - Nagoya City University West Medical Center, Aichi
  - Nagoya City University East Medical Center, Aichi
  - Naika Tonyobyonaika Maejima Iin, Aichi
  - Nagoya City University Hospital, Aichi
  - Tohno Chuo Clinic, Aichi
  - Kamagaya General Hospital, Chiba
  - Japan Community Health care Organization Funabashi Central Hospital, Chiba
  - International University of Health and Welfare Narita Hospital, Chiba
  - National Hospital Organization Fukuokahigashi Medical Center, Fukuoka
  - Fukuoka Kinen Hospital, Fukuoka
  - National Hospital Organization Takasaki General Medical Center, Gunma
  - Hiroshima Prefectural Hospital, Hiroshima
  - Japan Community Health care Organization Hokkaido Hospital, Hokkaido
  - National Hospital Organization Kanazawa Medical Center, Ishikawa
  - Sakaide City Hospital, Kagawa
  - Tenyoukai Central Hospital, Kagoshima
  - Kawasaki Rinko General Hospital, Kanagawa
  - Matsuba Clinic, Kanagawa
  - Maekawa Medical Clinic, Kanagawa
  - Tsuzuki Azuma Clinic Primary care and Rheumatology, Kanagawa
  - Mutsukawa Clinic Primary care and Gastroenterology, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - NHO Kumamoto Saishun Medical Center, Kumamoto
  - Sakura Jyuji Hospital, Sakurajyuji Medical Corporation, Kumamoto
  - Minami Nagano Clinic, Nagano
  - Japan Organization of Occupational Health and Safety Nagasaki Rosai Hospital, Nagasaki
  - Ikoma City Hospital, Nara
  - Nagaoka Chuo General Hospital, Niigata
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - Okayama University Hospital, Okayama
  - Tazuke Kofukai Medical Research Institute, Kitano Hospital, Osaka
  - Japan Community Health care Organization Osaka Minato Central Hospital, Osaka
  - Rinku General Medical Center, Osaka
  - Omi Medical Center, Shiga
  - Kuramochi Clinic Interpark, Tochigi
  - Tokyo center clinic, Tokyo
  - Tokyo Saiseikai Central Hospital, Tokyo
  - Kitasato University Kitasato Institute Hospital, Tokyo
  - Sumida General Clinic, Tokyo
  - Edogawa Hospital, Tokyo
  - Koto Hospital, Tokyo
  - Mishuku Hospital, Tokyo
  - Shimamura Memorial Hospital, Tokyo
  - Minamino Cardiovascular Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - Ome Municipal General Hospital, Tokyo
  - Toyama University Hospital, Toyama
  - Japan Organization of Occupational Health and Safety Toyama Rosai Hospital, Toyama
  - Toyama City Hospital, Toyama
  - Japan Organization of Occupational Health and Safety Wakayama Rosai Hospital, Wakayama
  - National Hospital Organization Minami Wakayama Medical Center, Wakayama
- Thailand (3):
  - Srinagarind Hospital, Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi
  - Ratchaburi Hospital, Ratchaburi Provinc

REFERENCES:
- [Result] Mikamo H, Takahashi S, Yamagishi Y, Hirakawa A, Harada T, Nagashima H, Noguchi C, Masuko K, Maekawa H, Kashii T, Ohbayashi H, Hosokawa S, Maejima K, Yamato M, Manosuthi W, Paiboonpol S, Suganami H, Tanigawa R, Kawamura H; IVERMILCO Study Group. Efficacy and safety of ivermectin in patients with mild COVID-19 in Japan and Thailand. J Infect Chemother. 2024 Jun;30(6):536-543. doi: 10.1016/j.jiac.2023.12.012. Epub 2023 Dec 27. PMID 38154616